CLINICAL TRIAL: NCT03368079
Title: Utilization of Negative Pressure Suction to Reduce Aspiration in Oropharyngeal Dysphagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 836211
Record Dates: First submitted 2017-10-29; First posted 2017-12-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Oropharyngeal Dysphagia
Keywords: Dysphagia; Oropharyngeal dysphagia; Video Fluoroscopic Swallowing Exam (VFSE)
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Negative Pressure Suction Device (Experimental)
  Interventions: Device: Negative Pressure Suction Catheter

INTERVENTIONS:
Device: Negative Pressure Suction Catheter — The negative pressure suction device to be used in the study will be a Foley catheter. The catheter will be placed through the gastrostomy tube site, directed retrograde through the esophagus, and terminating in the PES.

SUMMARY:
This is an investigator initiated prospective study to determine whether the use of a negative pressure suction in the hypopharynx will reduce the amount of aspiration during Video Fluoroscopic Swallowing Exam (VFSE) among patients with oropharyngeal dysphagia.

DETAILED DESCRIPTION:
During a properly coordinated swallow, the oropharynx, larynx, and hypopharynx undergo a series of movements that serve to prepare and expand the pharyngoesophageal segment (PES), which is the inlet into the esophagus. Under normal circumstances, a food bolus is safely propelled from the oropharynx, through the PES, and into the esophagus. Surgical and radiation therapy in the head and neck, as well as deficiencies such as poor coordination, mistiming, or obstructing lesions may prevent the food bolus from safely entering the esophagus and instead diverting toward the trachea.

A number of patients with severe oropharyngeal dysphagia are not able to tolerate any diet without risking aspiration and subsequent pneumonia, often to a degree severe enough that they cannot manage to safely swallow their secreted saliva. These patients depend on a gastrostomy feeding tube in order to obtain adequate daily nutritional requirements and must suction or spit out their saliva to prevent aspiration and a sensation of asphyxiation. Despite these precautions, many of these patients ultimately suffer life-threatening pneumonia. Investigators will be testing if the use of use of a negative pressure suction in the hypopharynx will reduce the amount of aspiration during Video Fluoroscopic Swallowing Exam (VFSE) among patients with severe oropharyngeal dysphagia

ELIGIBILITY:
Inclusion Criteria:

* Patients with videofluoroscopic evidence of aspiration with Rosenbek Penetration Aspiration Scale (PAS) greater than 5 for all tested food consistencies
* Gastrostomy tube dependence
* Exhaustion of conventional treatment options (physical, medical, and surgical therapies)

Exclusion Criteria:

* Complete PES stricture
* Inability to follow commands
* Current malignant disease
* No gastrostomy tube present
* Less than two years of cancer-free survival (if applicable)
* Vulnerable populations: adults unable to consent, pregnant women, and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Degree of aspiration | During VFSE, from the beginning of administration of the first bolus size to completion of the VFSE
  Degree of aspiration or laryngeal penetration, evaluated by the validated Rosenbek Penetration-Aspiration Scale (PAS). The PAS scale is an 8-point (1 to 8), equal-appearing interval scale:
  1. Material does not enter airway
  2. Material enters the airway, remains above the vocal folds, and is ejected from the airway.
  3. Material enters the airway, remains above the vocal folds, and is not ejected from the airway.
  4. Material enters the airway, contacts the vocal folds, and is ejected from the airway.
  5. Material enters the airway, contacts the vocal folds, and is not ejected from the airway.
  6. Material enters the ariway, passes below the vocal folds, and is ejected into the larynx or out of the airway.
  7. Material enters the airway, passes below the vocal folds, and is not ejected from the trachea despite effort.
  8. Material enters the airway, passes below the vocal folds, and no effort is made to eject.
Pharyngo-esophageal Segment (PES) opening size | During VFSE, PES is measured when the patient administers 20 cc of liquid barium and the PES is maximally distended.
  Pharyngo-esophageal Segment (PES) is a 2.5 to 4.5 cm manometric high-pressure zone located between the pharynx and esophagus. Normal Pharyngoesophageal segment opening size on lateral view: 0.80 cm +/- 0.40 cm

SECONDARY OUTCOMES:
Pharyngeal Constriction Ratio (PCR) | Measurement of the pharyngeal area during maximum contraction are taken after administration of 20 cc liquid barium. The pharyngeal area at rest is measured when 1 cc bolus is held in the oral cavity.
  Pharyngeal Constriction Ratio: is a measure of pharyngeal clearance pressure. It is calculated by dividing the lateral pharyngeal area during maximal contraction by the area with a 1 cc bolus held in the oral cavity. The area is determined by onscreen tool provided. Normal PCR: 0.14 +/- 0.28
Oropharyngeal transit time | Time from when bolus head first passes posterior nasal spine to time bolus head enters base of vallecula
  Oropharyngeal transit time is measured when the patient administers 20 cc of liquid barium. Normal oropharyngeal transit time: 0.42 sec +/- 0.36 sec
Hypopharyngeal transit time | Time from when bolus head exits the vallecula to time when bolus tale exits PES
  Hypopharyngeal transit time: is measured when the patient administers 20 cc of liquid barium. Normal Hypopharyngeal transit time: 0.77 sec +/- 0.26 sec

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-negative-pressure-suction-to-reduce-aspiration-inhaling-food-into-lungs-oropharyngeal-dysphagia-swallowing-disorder-672909/